CLINICAL TRIAL: NCT00890123
Title: Preoperative Intravenous Omega 3 Fatty Acids Administration in Elderly Patients Undergoing Hip Surgery: A Prospective, Randomized, Open-label, Comparative Clinical Trial
Brief Title: Preoperative Intravenous Omega 3 Fatty Acids Administration in Elderly Patients Undergoing Hip Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nizam's Institute of Medical Sciences University, India (Other)
Responsible Party: Principal Investigator, Dr. R. Gopinath, Professor, Nizam's Institute of Medical Sciences University, India
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NIMS/2008/Omegaven/Surgery/01
Record Dates: First submitted 2009-04-28; First posted 2009-04-29 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-10

CONDITIONS: Hip Surgery
Keywords: Omega 3 Fatty Acids; Inflammation; Hip Surgery; Inflammatory status; Infectious complications
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omegaven (Active Comparator): Patients in this arm will receive IV Omega 3 fatty acids (Omegaven®) for 3 days preoperatively.
  Interventions: Dietary Supplement: Omegaven-IV FO
- Without Omegaven (No Intervention): Patients will not receive IV Omega 3 fatty acids

INTERVENTIONS:
Dietary Supplement: Omegaven-IV FO — Will receive IV Omega 3 fatty acids (Omegaven®) for 3 pre operative days
  Arms: Omegaven

SUMMARY:
The perioperative administration of n-3 fatty acids has been shown to lead to favorable effects on outcome in patients with severe surgical interventions by lowering the magnitude of inflammatory response and by modulating the immune response. No study with preoperative administration of IV omega 3 fatty acids as a part of total parenteral nutrition (TPN) or monotherapy with it to demonstrate its effects on inflammatory and immune response has been conducted. So, this study has been planned to judge the inflammatory response of preoperative monotherapy with IV omega 3 fatty acids in elderly patients undergoing hip surgery considering the hyper-inflammation associated with this type of surgery in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

1. Elderly male or female patients undergoing hip surgeries
2. Age > 60 years
3. The patients who give written informed consent

Exclusion Criteria:

1. Refusal to participate in the study
2. Allergy to any of the constituents of nutritional products
3. HIV positive patients, patients with primary diagnosis of hypertriglyceridemia, patients on long term steroid therapy and cyclooxygenase inhibitors (more than 3 months)
4. Severe cardiac disease, hepatic disorders (total bilirubin > 1.5 times the upper limit of normal), psychiatric disorders likely to affect compliance, severe hemorrhagic disorders, stroke, embolism
5. Uncontrolled severe renal failure (Serum creatinine > 2 mg/dL) without dialysis/hemofiltration
6. Participation in any other clinical trial within the last 2 months

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-04; Primary Completion 2010-04 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
IL-6, 8, 10, HS-CRP levels | 5 days

SECONDARY OUTCOMES:
Infectious complications | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Dr R Gopinath, Principal Investigator — Professor and Head, Department of Anesthesia and critical care
Locations (1):
- Nizam's Institute of Medical Sciences, Hyderabad, Andhra Pradesh, India